CLINICAL TRIAL: NCT01884831
Title: Phase 2 The Use of Tissue-equivalent Based on Cultured Cells for Healing Skin Blemishes
Brief Title: The Study of the Effectiveness of Tissue Equivalent on the Basis of Cultured Cells to Heal Skin Blemishes
Acronym: SETES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ural State Medical University (Other)
Responsible Party: Principal Investigator, Korotkov Artem Vladimirovich, Senior Research Fellow, Ural State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: USMA01082012
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Neurotrophic Ulcers; Burns
Keywords: damage to the skin, the skin equivalent, cell therapy
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cell therapy (Experimental): study of the efficacy of skin equivalent comprising living cells and skin biodegradable substrate for the treatment of skin lesions
  Interventions: Biological: study of the efficacy of skin equivalent comprising living cells and skin biodegradable substrate for the treatment of skin lesions

INTERVENTIONS:
Biological: study of the efficacy of skin equivalent comprising living cells and skin biodegradable substrate for the treatment of skin lesions

SUMMARY:
In Russia the treatment nonhealing skin defects often limited to surgical interventions, despite having developed modern methods of treatment of non-healing ulcers and other skin imperfections. During the many years of research we have developed a skin equivalent comprising living cells.

During pilot trial showed that the skin equivalent provides healing skin defect within 1-4 weeks in 95% of patients.

ELIGIBILITY:
Inclusion Criteria:

* The presence of non-healing ulcer at least a month, an area of not less than 3 cm2 or smaller area of deep defects;
* Availability of burns II or III level;
* Epidermolysis bullosa;
* Availability of post-burn scars
* Defects in the skin after surgery

Exclusion Criteria:

* Acute and chronic diseases in the acute stage;
* Autoimmune diseases of connective tissue (collagen);
* Immunodeficiency states;
* System of inflammatory diseases of the skin;
* Conduct an aggressive corticosteroid therapy;
* Acute coronary syndrome;
* Acute disorders of cerebral circulation;
* Availability of local inflammation in the acute stage;
* Pregnancy;
* Breast-feeding.
* Positive results of the following tests: Anti-HIV-1 and -2, HIV-1Ag, anti-HTL VI and-II, anti-HbcorAg, HBs-Ag, anti-HCV, anti-CMV, anti-Toxoplasma gondii, RW, Neisseria gonorrheae, Chlamydia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
efficiency | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oleg G Makeev, MD, Study Chair — Ural State Medical University
Locations (1):
- Ural State Medical Academy, Yekaterinburg, Russia